CLINICAL TRIAL: NCT06806241
Title: Investigation of the Effects of Tranexamic Acid Solution Irrigation on Bleeding, Surgical Field Visibility, and Postoperative Edema in the Extraction of Horizontally Impacted Third Molars
Brief Title: Effects of Tranexamic Acid Irrigation on Impacted Third Molar Surgery
Status: Recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: E.142551
Record Dates: First submitted 2025-01-27; First posted 2025-02-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Bleeding; Tooth Extraction
Keywords: bleeding; tranexamic acid; wisdom teeth removal; edema
MeSH Terms: conditions — Hemorrhage; Edema | interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- saline irrigation group: In the double-blind, controlled, randomized study, only saline will be used as the irrigation solution in the control group patients.
  Interventions: Drug: saline irrigation
- tranexamic acid Irrigation group: In the double-blind, controlled, randomized study, saline with tranexamic acid solution will be used as the irrigation solution in the study group patients.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — in the study group, a combination of two ampules of Tranexamic acid solution mixed with saline will be used. Intraoperative bleeding, surgical field visibility, and postoperative edema will be monitored.
  Groups: tranexamic acid Irrigation group
Drug: saline irrigation — In control group, saline will be used for irrigation.Intraoperative bleeding, surgical field visibility, and postoperative edema will be monitored.
  Groups: saline irrigation group

SUMMARY:
Tranexamic acid (TXA) is an effective hemostatic agent used to reduce blood loss and the need for transfusion. It is a relatively safe drug with minimal significant side effects. The most commonly reported complications include nausea, diarrhea, and occasional orthostatic reactions. The increased risk of thromboembolic events associated with the drug is the most serious complication; however, this has not been reported in most clinical studies and remains uncertain. Based on experience from other types of surgeries, tranexamic acid appears to be safe for use without an increased risk of venous thrombosis. To mitigate systemic absorption and minimize undesirable side effects, TXA can be applied topically rather than intravenously, reducing the risk of venous thromboembolism.

DETAILED DESCRIPTION:
Topical TXA irrigation has recently begun to be used intraoperatively. In a study conducted by Eftekharian et al., the application of intraoperative 1% TXA irrigation solution during bimaxillary orthognathic surgery was found to be significantly associated with a reduction in intraoperative blood loss compared to placebo. Additionally, the topical application of TXA to the maxillary sinus during endoscopic sinus surgery has been shown to reduce intraoperative blood loss. In the current literature, the use of tranexamic acid irrigation during tooth extraction under local anesthesia has not been reported. Our study aims to demonstrate the effectiveness of TXA irrigation during the extraction of bone-retained teeth and its effect on postoperative edema.

ELIGIBILITY:
Inclusion Criteria:

1. Indicated for the Extraction of Bilaterally Impacted Third Molars with Bone Retention.
2. Systemically healthy patients aged 14-40 years with no bleeding disorders.

Exclusion Criteria:

1. Patients with systemic diseases affecting general health.
2. Patients diagnosed with any bleeding disorder.
3. Patients with advanced infection or cysts associated with the impacted tooth.

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
postoperative edema | 3 days
  Anatomical landmarks, including gonion (Go), ala nasi (AN), tragus (Tr), and lateral canthus (Ka), will be marked with methylene blue for measurement purposes.
  The distances between lateral canthus and gonion, tragus and commissure, and gonion and ala nasi will be measured preoperatively (just before the procedure begins) and on postoperative day 3, when maximum edema is expected, and the values will be recorded.

SECONDARY OUTCOMES:
intraoperative bleeding | during the surgery time
  During the surgery, the total aspirate volume collected in the suction device will be recorded. By subtracting the amount of irrigation solution used, the amount of bleeding (in cc) will be calculated separately for the right and left sides and documented.
intraoperative vision scale | during the surgery
  Intraoperatively, based on the evaluation of surgical bleeding and surgical comfort, the surgeon will be asked to rate the surgical field on a 5-point scale after irrigation. An average score will be calculated postoperatively to determine the surgical field evaluation score. Separate scoring will be performed for both the right and left sides.
  Scale:
  1. - Intense bleeding, making it impossible to isolate the tooth.
  2. - Severe bleeding, making isolation difficult.
  3. - Moderate bleeding, causing slight difficulty in isolation.
  4. - Mild bleeding, isolation is unaffected.
  5. - No bleeding or an almost bloodless surgical field.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Universty, Istanbul, Fatih, Turkey (Türkiye)